CLINICAL TRIAL: NCT02427776
Title: A Clinical Trial to Document Safety and Radiological Disease Activity in Patients With Relapsing-remitting Multiple Sclerosis Treated With Autologous CD4+ T Cells, Stimulated and Expanded ex Vivo by a Myelin Oligodendrocyte Glycoprotein Peptide Modified by the Introduction of a Thioreductase Motif Into the Flanking Residues of the Cell Epitope - A First-in-human Trial (SCLEROLYM TRIAL)
Brief Title: A Trial for Evaluating Both Safety and Preliminary Efficacy of a Single Infusion of Stimulated Autologous CD4+T Cells in Patients With Relapsing- Remitting Multiple Sclerosis
Acronym: SCLEROLYM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study ended prior enrollment of the first patient because of unexpected issues in the manufacturing process prevented production of adequate clinical batches
Sponsor: Imcyse SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS/MOGMOD/CT/FIH/01
Record Dates: First submitted 2015-04-02; First posted 2015-04-28 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMP (Experimental)
  Interventions: Biological: Autologous CD4+T cells stimulated and expanded ex vivo by a MOG peptide modified by the introduction of a thioreductase motif into the flanking residues of the T cell epitope

INTERVENTIONS:
Biological: Autologous CD4+T cells stimulated and expanded ex vivo by a MOG peptide modified by the introduction of a thioreductase motif into the flanking residues of the T cell epitope — 1 administration comprising 5 - 50 millions of cells

SUMMARY:
The purpose of this study is to assess the safety and the preliminary efficacy of a single infusion of stimulated autologous CD4+ T cells in patients with Relapsing-Remitting Multiple Sclerosis.

The study duration for the patients (from start of baseline to end of follow-up) is 270 days.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 60 years of age
* Patients closely followed up for at least one year prior to inclusion (i.e. prior to the start of the baseline phase) if the diagnosis of the disease was made more than one year ago, to ensure that all possible episodes of clinical relapses which occurred during this interval of time were recorded and documented
* Multiple sclerosis that meets the 2010 revised McDonald criteria
* Relapsing/remitting type of multiple sclerosis (which includes clinically isolated syndromes if imaging shows brain lesions disseminated in space and time)
* Radiologically active disease defined by at least one gadolinium-enhancing lesion on a T1-weighted magnetic resonance imaging brain scan performed recently (i.e. within 3 months prior to inclusion)
* Disease-modifying drug naïve patients or patients with stable and adequately taken disease-modifying therapy (interferon β-1, glatiramer acetate, or dimethyl fumarate) for at least six months before inclusion (NOTE: Other disease modifying drugs might be added at a later date, depending on the results of current investigations)
* EDSS Score <= 5.5
* Positive predictive test in vitro for patient's CD4+ cell reactivity to immunogenic peptide
* Women of childbearing age must have a negative pregnancy test and must use adequate contraception during the treatment and follow-up phase of the study (three pregnancy tests will be required prior to and during the study: (1) during the screening phase, (2) about one week prior to leukapheresis, and (3) about one week prior to re-infusion of autologous cells)
* Fully informed written consent obtained

Exclusion Criteria:

* Positive only for the HLA DRB1*0101, DRB1*0102, DRB1*0401, DRB1*0426 alleles or for the combination of the previous alleles.
* Evidence of clinical relapse and use of intravenous or oral corticosteroids within 30 days prior to inclusion
* Therapeutic escalation anticipated (including change of disease modifying drug), other than the cell-based immunotherapy of this study, within the next six months
* Significant coexisting systemic disease including renal insufficiency
* Positive serology for hepatitis B and C, AIDS and syphilis
* Participation in another interventional clinical study, currently or during the past three months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Safety of the cell based immunotherapy (Adverse events) | 6 months
  Adverse events
Safety of the cell based immunotherapy (Vital signs) | 6 hours
  Vital signs
Safety of the cell based immunotherapy (Physical examination) | 6 months
  Physical examination
Safety of the cell based immunotherapy (Laboratory parameters) | 6 months
  Laboratory parameters
Safety of the cell based immunotherapy (MRI) | 6 months
  MRI

SECONDARY OUTCOMES:
MRI derived parameters | 3 months before the day of administration of the investigational medicinal product, the day of administration, 45, 90, 135 and 180 days after the administration
  * Cumulative number and mean number per scan of active inflammatory lesions
  * Cumulative number and mean number per scan of new lesions
  * Cumulative number and mean number per scan of enlarged lesions
Expanded Disability Status Scale (EDSS) | 3 months before the day of administration of the investigational medicinal product, the day of administration, 45, 90, 135 and 180 days after the administration
Clinical relapses | 3 months before the day of administration of the investigational medicinal product, the day of administration, 45, 90, 135 and 180 days after the administration
Circulating MOG specific cytolytic CD4+ cells | 3 months before the day of administration of the investigational medicinal product, the day of administration, 45, 90, 135 and 180 days after the administration
Circulating anti-MOG antibodies | 3 months before the day of administration of the investigational medicinal product, the day of administration, 45, 90, 135 and 180 days after the administration

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels
  - University Hospital Leuven (Gasthuisberg), Leuven
  - University Hospital of Liège, Liège